CLINICAL TRIAL: NCT04092842
Title: Evaluation of a New Technique to Fill the Defect Generated After Conservative Surgery in Breast Cancer: Randomized Clinical Trial
Brief Title: Evaluation of a New Technique to Fill the Defect Generated After Conservative Surgery in Breast Cancer
Acronym: PROSILMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-SIL-2017-70
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Breast Conserving Surgery
Keywords: Breast Neoplasms; Breast Conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Group whith silicone prothesis Group whith standard surgical procedure
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group intervention: Silicone prothesis (Experimental): Breast cancer conservative surgery will be performed by removing the tumor according to the usual technique and then the defect generated will be filled with a silicone prosthesis of the same size. Said prosthesis will be covered with fat and subcutaneous cellular tissue and then the skin will be closed.
  Interventions: Device: Silicone prosthesis
- Group control: Usual surgical technique (Active Comparator): Breast cancer conservative surgery will be performed according to the usual surgical technique, that is, removing the tumor and covering the defect by mobilizing the breast tissue and then closing the skin.
  Interventions: Procedure: Usual practice

INTERVENTIONS:
Device: Silicone prosthesis — Silicone prosthesis
  Arms: Group intervention: Silicone prothesis
Procedure: Usual practice — Usual surgery
  Arms: Group control: Usual surgical technique

SUMMARY:
The placement of a small silicone prosthesis in the partial defects generated by conservative breast cancer surgery improves the aesthetic result, compared to the usual surgical technique, in a safe and reproducible way and compatible with adjuvant treatments. It could also potentially improve the quality of life of patients

DETAILED DESCRIPTION:
Conservative surgery in breast cancer is performed more than 50% of cases, however, aesthetic results are suboptimal, because reconstructive techniques are performed in less than 5% of them. Objective: To demonstrate that the placement of a silicone prosthesis in partial defects generated by breast cancer conservative surgery improves the aesthetic result, compared to the usual surgical technique, safely, reproducibly and compatible with adjuvant treatments.

Methodology: Prospective randomized clinical trial, controlled with blind evaluator. Inclusion criteria: Women with breast cancer candidates for conservative surgery. Intervention: In the cases the study technique will be carried out consisting in the filling of the defect with a silicone prosthesis of size adjusted to it (2-4cm). Controls: usual surgical procedure. Main result variable: aesthetic results (visual analog scale) according to the patient, surgeon and blind external evaluator. Secondary variables: surgical complications, local complications derived from adjuvant treatments, rate of local recurrence, rate of reintervention due to affected margins, behavior in mammographic follow-up, professional satisfaction and impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

- Women, over 18 years old, with breast cancer who attend breast pathology consultations at the Sant Pau Hospital in which conservative surgery is indicated.

Exclusion Criteria:

* Multicentric tumors
* Tumors larger than 5cm
* Locally advanced tumors (T4): Deep plane involvement or skin involvement
* Patients in stages IV (distance dissemination)
* Patients who need mastectomy
* Patients with disabilities or who do not understand the terms of the study or do not agree to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Aesthetic result | 4 weeks
  Aesthetic result of the new technique by applying a visual analog scale for measuring patient satisfaction.
  Scale ranges: minimum score: 0 (no satisfaction - worse outcome), maximum score: 10 (total satisfaction - better outcome)

SECONDARY OUTCOMES:
Surgical complications | 4 weeks
  Incidence of surgical complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain